CLINICAL TRIAL: NCT03721393
Title: Data Collection - Of Syncope Tilt Table Testing Study
Acronym: COST3
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C2109
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Orthostatic Hypotension; Reflex Syncope
Keywords: tilt table test, valsalva
MeSH Terms: conditions — Hypotension, Orthostatic; Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Syncope patients: Patients that have undergone an ARS assessment and diagnosed with orthostatic hypotension or reflex syncope.
  Interventions: Device: Wearable heart monitor
- Group 2: Control patients: Patients that have undergone an ARS assessment and are control subjects.
  Interventions: Device: Wearable heart monitor

INTERVENTIONS:
Device: Wearable heart monitor — Participants will be fitted with a wearable heart monitor placed on the skin that measures physiologic signals. There is no intervention or treatment.

SUMMARY:
To characterize the impact of orthostatic hypotension (OH) and reflex syncope on signals measured using a wearable cardiac monitor prototype device.

To evaluate the relationship of signals measured from the wearable cardiac monitor prototype device with reported symptom severity of orthostatic intolerance per standard data collection, analysis, and questionnaires.

DETAILED DESCRIPTION:
This is a non-randomized feasibility study that will enroll up to 50 participants that have undergone a previous autonomic reflect screen (ARS) assessment and were either diagnosed with OH or reflex syncope, or considered to be control subjects for this study.

A maximum of 20 subjects diagnosed with reflex syncope, a maximum of 10 subjects diagnosed with OH and a maximum of 10 control subjects will be enrolled. There will be one study visit per subject.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to provide informed consent
* Age 18 or above
* No contraindications to undergo tilt table test, Valsalva maneuver test, and deep breathing test (Components of the ARS assessment)
* Previously underwent a clinically indicated ARS assessment without complications (including deep breathing, Valsalva maneuver, and tilt table testing). Previously diagnosed with OH, reflex syncope, OR control subjects assessed as normal, based on the ARS assessment. Patient enrollment shall be based on the type of diagnosis.
* Willing to participate in one additional tilt table test, Valsalva maneuver test, and deep breathing test (components of the ARS assessment)

Exclusion Criteria:

* Currently enrolled in another clinical trial that might interfere with data collection.
* Subject is pregnant or planning to become pregnant during the study
* Active Implantable Medical Device, e.g. cardiac implantable electronic devices, bladder stimulators, diaphragm stimulators, implantable neuro stimulator, implantable active monitoring devices, implantable active drug administration devices, etc.
* Have a prosthetic cardiac valve or previously underwent cardiac valve surgery.
* Known allergy to materials used in the study (adhesive, ECG electrodes)
* Diagnosed with syncope due to cardiologic causes.
* Have had a myocardial infarction in the previous 90 days
* Have been diagnosed with tachycardia that requires medical treatment
* Experienced complications during previous clinically indicated ARS assessment
* Are on medications that could affect autonomic function, if considered not safe or unwilling to hold such medications for at least four half-lives prior to testing (judged by the study Principal Investigator)
* Have any contraindication for tilt test, Valsalva maneuver test or deep breathing test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have previously undergone a ARS assessment and were diagnosed with OH or reflex syncope, or are control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Physiologic Signal Detection | 12 months
  Characterize the impact of orthostatic hypotension (OH) and reflex syncope on physiologic signals measured using a wearable cardiac monitor prototype device.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Singer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Foundation, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No